CLINICAL TRIAL: NCT00228397
Title: A Multicenter, Randomized, Double-blind, Long-term Extension Study to Determine the Safety, Tolerability, and Preliminary Efficacy of CCI-779 in Subjects With Relapsing Multiple Sclerosis.
Brief Title: Study Evaluating CCI-779 in Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3066A2-210
Record Dates: First submitted 2005-09-16; First posted 2005-09-28 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — temsirolimus

INTERVENTIONS:
Drug: CCI-779

SUMMARY:
To evaluate the safety and tolerability of long-term therapy with 3 dose levels of oral CCI-779 administered to subjects with relapsing MS who completed study 3066A2-205-WW.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with relapsing-remitting MS or secondary progressive MS with relapses.
* Successful completion of study 3066A2-205-WW with no major protocol violations.

Exclusion Criteria:

* Pregnancy or lactation.
* Clinically important abnormalities on the physical examination, vital signs, or electrocardiogram (ECG) performed at the last visit of study 3066A2-205-WW (day 252).
* Any adverse events or findings observed in study 3066A2-205-WW that in the opinion of the investigators would preclude the subject's entry into the extension study.

Please refer to section 16.2 'Discontinuation and Withdrawal of Subjects' regarding withdrawal of patients who have any clinical abnormalities in hematology or laboratory test results obtained at the last visit of the double-blind active phase of study 3066A2-205-WW.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2003-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Long-term safety.
Listing and summary tables of AE and TEAEs, vital signs, laboratory evaluations, and ECG data will be generated.

SECONDARY OUTCOMES:
Preliminary efficacy of long-term treatment.
Lesions observed on MRI scans, clinical measures such as the EDSS scale, the 9-Hole Peg Test, the Paced Auditory Serial Addition Test and the Timed Ambulation 25-Foot Test, occurrence of relapse, will be analyzed at end -point (12 or 16 months).
Only descriptive statistics will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer